CLINICAL TRIAL: NCT00999492
Title: Selection of Aspheric Diffractive Multifocal IOLS Based on Corneal Wavefront
Brief Title: Selection of Aspheric Diffractive Multifocal Intraocular Lens (IOLS) Based on Corneal Wavefront
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mark Packer, MD, FACS (Other)
Responsible Party: Sponsor-Investigator, Mark Packer, MD, FACS, Sponsor-Investigator, Drs. Fine, Hoffman and Packer, LLC
Organization: Drs. Fine, Hoffman and Packer, LLC (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMF-09-001; NCT01061892 (obsolete NCT alias)
Record Dates: First submitted 2009-10-19; First posted 2009-10-21 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Cataracts
Keywords: Tecnis Multifocal; Patients scheduled for cataract or lens replacement surgery with implantation of multifocal intraocular lenses
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Tecnis® Multifocal (TMF) — Aspheric, diffractive multifocal intraocular lenses

SUMMARY:
Given the availability of aspheric diffractive IOLs with varying negative spherical aberration it may be feasible, by selecting the best fit IOL, to minimize aberrations and thereby maximize visual performance.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Scheduled to undergo bilateral cataract or refractive lens surgery
* Visual potential of 20/30 or better in each eye after lens removal and IOL implantation
* Naturally dilated pupil size (in dim light) > 3.5 mm (with no dilation medications) for both eyes
* Preoperative regular corneal astigmatism of 2.5 D or less
* Clear intraocular media other than cataract
* Availability, willingness, and sufficient cognitive awareness to comply with examination procedures

Exclusion Criteria:

* Ocular disease other than cataract which could potentially limit uncorrected visual acuity or visual performance.
* Astigmatism not correctable by limbal relaxing incisions (greater than 2.5 D)
* Use of systemic or ocular medications that may affect visual outcomes
* Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus, immunocompromised, etc.)
* Uncontrolled systemic or ocular disease
* History of ocular trauma or prior ocular surgery
* Amblyopia or strabismus
* Known pathology that may affect visual acuity; particularly retinal changes that affect vision (macular degeneration, cystoid macular edema, proliferative diabetic retinopathy, etc.)
* Diagnosed degenerative visual disorders (e.g. macular degeneration, or other retinal disorders) that are predicted to cause future acuity losses to a level of worse than 20/30
* Subjects who may be expected to require retinal laser treatment or other surgical intervention
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome)
* Pupil abnormalities (non-reactive, tonic pupils or abnormally shaped pupils)
* Contact lens usage within 6 months for PMMA lenses, 1 month for gas permeable lenses or 1 week for extended-wear and daily-wear soft lenses
* Requiring an intraocular lens power <15.0 or >26.0 diopters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Frequency of spectacle wear | 3 months postoperatively

SECONDARY OUTCOMES:
Frequency and degree of visual symptoms | 3 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Drs. Fine, Hoffman and Packer, LLC, Eugene, Oregon, United States